CLINICAL TRIAL: NCT02726906
Title: Lifestyle Enriching Activities for Research in Neuroscience Intervention Trial: LEARNit Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Judy Pa, Assistant Professor of Neurology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG046928
Record Dates: First submitted 2016-03-28; First posted 2016-04-04 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Aging; Cognitive Ability, General
Keywords: Alzheimer's disease; Mild Cognitive Impairment; Brain Imaging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate-aerobic walking (Experimental): Participants will complete a 6-month home-based moderate-aerobic walking program of 150 minutes per week with the assistance of an interventionist.
  Interventions: Behavioral: Moderate-aerobic walking; Radiation: Positron Emission Tomography (PET) scan; Device: Physical activity monitor
- Healthy Living Education (Placebo Comparator): Participants will receive monthly topics on healthy living lifestyles for self-paced reading over 6 months with the assistance of an interventionist.
  Interventions: Radiation: Positron Emission Tomography (PET) scan; Behavioral: Healthy living education; Device: Physical activity monitor

INTERVENTIONS:
Behavioral: Moderate-aerobic walking
  Arms: Moderate-aerobic walking
Radiation: Positron Emission Tomography (PET) scan — Radioligand that binds to proteins using a PET/CT scanner.
Behavioral: Healthy living education
  Arms: Healthy Living Education
Device: Physical activity monitor — Wrist device that will track daily physical activity

SUMMARY:
The purpose of this study is to examine the effects of modifiable lifestyle factors including exercise and healthy living on brain health. The investigators will compare 2 types of interventions, moderate aerobic walking vs. healthy living education, over 6 months to evaluate changes in brain health, cognition, and physical function in older adults with cognitive concerns.

DETAILED DESCRIPTION:
Cognitive decline in older adults is a major public health issue. The cost of caring for older adults with substantial cognitive impairment, like those with Alzheimer's Disease in the US is approximately $200 billion a year, causing major societal, economic, and caregiving burden. Despite great advances towards diagnosing these problems, the discovery of effective treatments has been minimal. Exploring non-pharmacological interventions, such as exercise and healthy living, have gained momentum. These promising, modifiable lifestyle interventions have the potential for delaying disease onset and slowing decline in cognition. However, the therapeutic effect of lifestyle interventions in patients with mild cognitive impairment, a prime intervention period for treatment, is not well understood. Therefore, in this study, the investigators will examine brain, body, and cognitive changes in older adults who engage in moderate-aerobic walking or healthy living education.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. English-speaking
3. 55-80 years old
4. Exhibits sedentary behavior
5. Objective cognitive impairment
6. Mini-Mental State Exam score > 26
7. Perform at least 1 standard deviations below normative values on cognitive tests
8. Absence of dementia
9. Ability to complete both MRI and PET scans
10. Physically capable of completing health programs

Exclusion Criteria:

1. Baseline dementia
2. History of a neurological disorder
3. Current psychiatric illness
4. Head trauma with a loss of consciousness > 10 minutes
5. Severe sensory deficits
6. Substance abuse
7. Depression (GDS < 8 of 15)
8. Inability to perform intervention (e.g., inability to walk without assistance)
9. Contraindications to MRI scan (e.g., pacemaker)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-08-21 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All data requests will be reviewed by the data committee. Approved investigators will be provided de-identified participant-level data from the trial as a .CSV file.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available starting July 1, 2025 and for at least 3 years.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants complete a 30-day run-in and baseline visit prior to randomization.
Groups:
- Moderate-aerobic Walking: Participants will complete a 6-month home-based moderate-aerobic walking program of 150 minutes per week with the assistance of an interventionist.
  Moderate-aerobic walking
  Positron Emission Tomography (PET) scan: Radioligand that binds to proteins using a PET/CT scanner.
  Physical activity monitor: Wrist device that will track daily physical activity
- Healthy Living Education: Participants will receive monthly topics on healthy living lifestyles for self-paced reading over 6 months with the assistance of an interventionist.
  Positron Emission Tomography (PET) scan: Radioligand that binds to proteins using a PET/CT scanner.
  Healthy living education
  Physical activity monitor: Wrist device that will track daily physical activity
Period: Overall Study
Arm/Group | Moderate-aerobic Walking | Healthy Living Education
Started | 33 | 33
Completed | 30 | 30
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate-aerobic Walking | Healthy Living Education | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.1) | 67.3 (6.4) | 67.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 26 | 31 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 24 | 26 | 50
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Brain Scan as a Measure of Brain Function
Description: Functional MRI has proven to be an effective non-invasive, in-vivo tool for measuring brain function via the BOLD signal. Growing evidence supports that fMRI BOLD can detect neuronal changes that occur very early in the disease process. The hippocampus has been shown to be a selectively vulnerable region in AD, and several studies, including our own, identified a aberrant brain signal in the hippocampus in older adults. The typical range for this outcome is -10 to 10 with higher scores indicating better brain function.
Time Frame: Baseline and Follow-up at 6 months
Population: Definition of ITT analysis sample: all eligible participants who (1) began the intervention and (2) completed baseline assessment and 6-month assessment for the primary analysis of fMRI BOLD and MST behavioral test. All consented, randomized participants are grouped according to the treatment assigned at randomization. MRI data was not available for one participant in the Healthy Living Education group, resulting in an N of 29 for all fMRI measures.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Moderate-aerobic Walking | Healthy Living Education
Number analyzed (Participants) | 30 | 29
units on a scale
  Baseline | -0.442 [-0.879 to -0.005] | -0.203 [-0.650 to 0.243]
  Follow-up | 0.018 [-0.274 to 0.310] | 0.033 [-0.267 to 0.333]

2. Primary Outcome: Mnemonic Similarity Test as a Measure of Memory (Cognition)
Description: The participants will encode a series of objects presented on a computer. Following the encoding period, they will begin their fMRI scan and be asked to indicate if they recognize the objects on the screen, which include targets (previously seen objects), lures (objects that are similar to previously seen objects) and novel (unrelated objects). The discrimination between Targets and Lures will indicate the rate at which participants "correctly reject" the Lures (via pattern separation) or "false alarm" to the Lures (via pattern completion). The theoretical range for this outcome is -1 to 1 with higher scores indicating better memory function.
Time Frame: Baseline and Follow-up at 6 months
Population: Definition of ITT analysis sample: all eligible participants who (1) began the intervention and (2) completed baseline assessment and 6-month assessment for the primary analysis of fMRI BOLD and MST behavioral test. All consented, randomized participants are grouped according to the treatment assigned at randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moderate-aerobic Walking | Healthy Living Education
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 0.32 [0.23 to 0.41] | 0.32 [0.23 to 0.41]
  Follow-up | 0.28 [0.18 to 0.37] | 0.36 [0.27 to 0.45]

3. Secondary Outcome: Amyloid Positron Emission Tomography (PET) Scan as a Measure of Tracer Binding (SUVr)
Description: Each participant received PET scans with Neuraceq [florbetaben F 18 (FBB)] to measure amyloid-beta PET binding. IV injections of the tracers (FBB, -8.11 6 0.6 mCi) were done outside of the scanning room. Four 5-min frames were acquired 90 minutes after injection.
Time Frame: Baseline and Follow-up at 6 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: standardized uptake value ratio (SUVr)
Arm/Group | Moderate-aerobic Walking | Healthy Living Education
Number analyzed (Participants) | 30 | 30
standardized uptake value ratio (SUVr)
  Baseline | 1.05 [0.99 to 1.11] | 1.01 [0.94 to 1.07]
  Follow-up | 1.05 [0.99 to 1.12] | 1.01 [0.94 to 1.08]

4. Secondary Outcome: Single-stage Treadmill Test
Description: This is a measure of cardiovascular fitness. This test has been validated against peak VO2 max with r=0.96. Heart rate response is monitored with a Polar heart rate monitor and the heart rate at the end of the 4 min test is used to estimate VO2max using an established equation for conversion. The theoretical range for this outcome is 0 to 200 with higher scores indicating better cardiovascular fitness.
Time Frame: Baseline and Follow-up at 6 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Moderate-aerobic Walking | Healthy Living Education
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 29.5 [27.4 to 31.6] | 30.0 [27.8 to 32.1]
  Follow-up | 31.2 [29.2 to 33.3] | 31.1 [29.0 to 33.2]

5. Secondary Outcome: Modified Physical Function Test
Description: This test is a measure of multiple domains related to functional activities of daily living. Each physical activity in score is of varying difficulty level. The theoretical range for this outcome is 0 to 36 with higher scores indicating better physical function.
Time Frame: Baseline and Follow-up at 6 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moderate-aerobic Walking | Healthy Living Education
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 33.1 [32.2 to 33.9] | 33.0 [32.1 to 33.9]
  Follow-up | 33.6 [32.7 to 34.4] | 33.7 [32.8 to 34.6]

6. Secondary Outcome: Brain-derived Neurotropic Factor (BDNF) as a Measure From Blood
Description: We will quantitatively analyze pre- and post-measurements of brain derived neurotrophic factor (BDNF). BDNF has been shown to increase after exercise intervention in humans and peripheral increases in these hormones correlate to cell proliferation in the dentate gyrus of the hippocampus. We measure total BDNF from plasma.
Time Frame: Baseline and Follow-up at 6 months
Population: Definition of ITT analysis sample: all eligible participants who (1) began the intervention and (2) completed baseline assessment and 6-month assessment for the primary analysis of fMRI BOLD and MST behavioral test. All consented, randomized participants are grouped according to the treatment assigned at randomization. BDNF Plasma sample for one participant in the Healthy Living Education group did not pass QC thresholds and was excluded from analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Moderate-aerobic Walking | Healthy Living Education
Number analyzed (Participants) | 30 | 29
pg/mL
  Baseline | 5.80 [3.13 to 8.46] | 8.11 [5.39 to 10.83]
  Follow-up | 6.15 [3.50 to 8.80] | 6.63 [3.87 to 9.39]

ADVERSE EVENTS:
Time Frame: Time between baseline and followup visit of 6-8 month intervention.
Arm/Group | Moderate-aerobic Walking | Healthy Living Education
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 11/30 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate-aerobic Walking (N=30) | Healthy Living Education (N=30)
Cardiac disorders (Cardiac disorders) | 1 | 0 — myocardial infarction, subsequent stent placement
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate-aerobic Walking (N=30) | Healthy Living Education (N=30)
Skin (Skin and subcutaneous tissue disorders) | 8 | 6 — Pain at injection site for PET scan tracer [12]; skin irritation due to cleaning agent for wearable device (accelerometer) [1], ankle swelling
Non-Hodgkins lymphoma (Blood and lymphatic system disorders) | 1 | 0
Falls (Musculoskeletal and connective tissue disorders) | 2 | 0 — One slipped on driveway, one slipped walking to car after a hike

LIMITATIONS AND CAVEATS:
Our study experienced delays due to the Covid-19 pandemic and impact on research. The human subjects portions of the trial were paused from March 2020 to August 2020 (a 5-month period of no human research activities on campus) due to local university Covid-19 restrictions. Once the pause was lifted, we were able to resume normal day to day activities with precautions in place, and have since completed the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT02726906/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT02726906/SAP_001.pdf